CLINICAL TRIAL: NCT04644744
Title: End-ischemic Hypothermic Oxygenated (HOPE) vs. Normothermic Machine Perfusion (NMP) Compared to Conventional Cold Storage in Donation After Brain Death Liver Transplantation; a Prospective Multicentre Randomized Controlled Trial (HOPE-NMP)
Brief Title: Hypothermic Oxygenated (HOPE) Versus Normothermic Machine Perfusion (NMP) in Human Liver Transplantation
Acronym: HOPE-NMP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Georg Lurje, MD, Consultant HPB- and Transplant Surgeon, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EA2/270/20
Record Dates: First submitted 2020-11-13; First posted 2020-11-25 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Hepatocellular Injury; Liver Transplant Disorder
Keywords: ex-vivo machine Perfusion; Hypothermic oxygenated machine perfusion; Normothermic machine perfusion; Orthotopic liver transplantation; Extended criteria donation; Donation after brain death; HOPE; NMP

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hypothermic oxygenated perfusion (HOPE) (Experimental): Application of end-ischemic Hypothermic machine perfusion (HOPE) for a minimum of 2 hours (until hepatectomy)
  Interventions: Device: Hypothermic oxygenated perfusion (HOPE)
- Normothermic machine perfusion (NMP) (Experimental): Application of end-ischemic normothermic machine perfusion (NMP) for a minimum of 4 hours (up to 24 hours)
  Interventions: Device: Normothermic machine perfusion (NMP)
- Conventional cold storage (CCS) (Active Comparator): Conventional cold storage
  Interventions: Device: Hypothermic oxygenated perfusion (HOPE); Device: Normothermic machine perfusion (NMP)

INTERVENTIONS:
Device: Hypothermic oxygenated perfusion (HOPE) — HOPE for 1 hour via the portal vein in a recirculating and pressure controlled system (2-3 mm Hg), 0.1 ml/g liver/min, perfusion volume 3-4 L, Belzer (UW) machine perfusion solution, perfusate temperature 10 °C, perfusate oxygenation pO2 of 60-80 kPa
  Other Names: Hypothermic machine perfusion (HMP)
  Arms: Conventional cold storage (CCS); Hypothermic oxygenated perfusion (HOPE)
Device: Normothermic machine perfusion (NMP) — End-ischemic NMP will be continued throughout the recipient hepatectomy and until the transplanting team is ready to implant the liver. The minimum protocol-stipulated NMP duration is 4 hours, the time needed for ATP repletion in animal studies. Total NMP preservation time will be according to the official recommendations of the manufacturer (4-24 hours) and at the discretion of the local transplant centre. The liver allograft will be disconnected from the OrganOx metra® device immediately prior to transplantation and flushed with three litres of HTK via the hepatic artery and the portal vein.
  Arms: Conventional cold storage (CCS); Normothermic machine perfusion (NMP)

SUMMARY:
The common practice of conventional cold storage (CCS) organ preservation has changed little since the initial introduction of the original University of Wisconsin (UW) organ preservation solution in the late 1980s. CCS relies on hypothermia to decelerate metabolism and reduce oxygen demand in order to prolong the time of ischemia without rapid functional graft impairment, therefore merely delaying graft damage. While CCS only prolongs storage time and limits the damage sustained during the period of cold ischemia, ex-vivo machine perfusion (MP) appears to be capable of reversing some of these effects. Currently, two main paradigms prevail in the clinical approach to liver allograft MP: hypothermic oxygenated MP (HOPE) may be seen as a dynamic alternative of the traditional organ preservation based on hypothermia-induced deceleration of metabolism, which aims to combine the positive effects of hypothermia observed in classical cold storage (e.g. technical simplicity, relative safety, decreased metabolism) with the positive effects of dynamic preservation (e.g. controlled sheer stress mediated gene activation, removal of metabolites, transport of oxygen and ATP recharging). Normothermic perfusion (NMP) aims at re-equilibration of cellular metabolism by preserving the organ at physiological temperatures whilst ensuring sufficient oxygen and nutrient supply. In both approaches, the perpetual circulation and moderate shear-stress sustain endothelial functionality. While past and current clinical trials were designed to compare different MP approaches with CCS as the clinical standard, a direct comparison between different end-ischemic MP techniques (HOPE versus NMP) is still lacking. The purpose of this study is to test the effects of end-ischemic NMP versus end-ischemic HOPE technique in a multicentre prospective randomized controlled clinical trial (RCT) on ECD liver grafts in DBD liver-transplantation (HOPE-NMP). Two-hundred-thirteen (n = 213) human whole organ liver grafts will be submitted to either 4-24 hours of NMP (n = 85) or 2-3 hours of HOPE (n = 85) directly before implantation and going to be compared to a control-group of patients (n = 43) transplanted with static cold storage preserved ECD-allografts. Primary (surgical complications as assessed by the comprehensive complication index [CCI]) and secondary (among others laboratory values, graft- and patient survival, hospital costs, hospital stay) endpoints are going to be analysed.)

DETAILED DESCRIPTION:
Liver transplantation has evolved as the mainstay of treatment for end-stage liver disease. While the demand for organ transplantation has increased over time, Germany's organ donation rate is low compared to other countries. The main indications for listing are 'fibrosis and cirrhosis' (27%) followed by 'alcoholic liver disease' (23%) and 'hepatic malignancies' (17%).

With the advent of emerging waiting list mortality, several strategies for donor pool expansion are being pursued; these include the use of living donors, splitting of cadaveric livers for two recipients, and the use of extended criteria donor (ECD) allografts for OLT. These ECD-allografts, however, exhibit poor tolerance to ischemia-reperfusion (I/R) injury, an important cause of liver damage. As such, I/R-injury is the underlying cause of graft dysfunction in ECD-allografts and negatively affects the process of liver regeneration in surgical conditions including hepatic resections and OLT.

Machine perfusion with oxygenated blood was already implemented in the first series of 11 successful human OLTs in the 1960s. While the logistical simplicity and reliable performance of CCS led to its quick adoption as the standard solid organ preservation technique, the increased utilization of high-risk organs has unveiled the limitations of CCS, furthering the debate on the impact of different MP techniques. Today, perfusion conditions vary broadly, especially in preclinical research. Parameters under discussion include different temperatures, perfusate composition, the application of perfusion flow (continuous or pulsatile), the timing and duration of the perfusion, starting either at the donor site or applied only end-ischemic in the recipient centre. Two main principles have been translated into clinical practice today: hypothermic oxygenated perfusion (HOPE) and normothermic MP (NMP). The latter differs significantly from HOPE because the allograft is perfused with oxygenated red blood cells or oxygen carriers at physiological temperatures with the aim to reduce the ischemic graft injury by minimizing the duration of cold preservation and perfectly mimicking physiological conditions. A recently completed randomized controlled trial (RCT) by Nasralla et al. proved the feasibility of NMP for OLT and demonstrated a significant reduction in peak AST and subsequent early allograft dysfunction (EAD), however without a significant difference in graft and patient survival. Most recently, a development of the NMP technique that allowed a 7-day preservation of human livers with a sustained metabolic function and an intact liver structure was recently reported by Eshmuminov et al. Based on the sustained full hepatic metabolism during NMP, several groups are currently exploring the possibility of normothermic viability testing. The cellular mechanisms of organ protection by NMP do not center around IRI mitigation and reconditioning, but IRI prevention, and are altogether different from cold perfusion techniques. While normothermic machine perfusion is most effective when applied during the entire period of organ preservation, the end-ischemic application of this technique in the recipient hospital is becoming more popular.

There are two main hypotheses on the underlying mechanisms of HOPE induced organ protection; (I.) modulation of cellular metabolism (energy household, mitochondrial respiration), and (II.) stimulation of the sinusoidal endothelial layer. Although, tissue oxygen consumption is markedly decreased at 4-10 Celsius, it is not completely suspended. The shift of mitochondrial metabolism to anaerobic pathways leads to expressed mitochondrial metabolite accumulation during ischemia and subsequently to extreme radical oxygen species (ROS) generation through rapid re-oxidization by the early reperfusion respiratory burst. The delivery of oxygen during cold preservation can effectively upload cellular energy household via various mitochondrial pathways. Pre-implantation resuscitation of organs with machine perfusion and oxygen can increase tissue ATP levels and decrease the post-ischemic production of ROS and danger-associated molecular patterns (DAMPs), this subsequently leads to a mitigated immune response. This organ conditioning effect is attributed to a controlled re-oxygenation inducing moderate ROS release just before reperfusion. These low levels of ROS are not only responsible for the induction of antioxidant enzymes (heme-oxygenase, gluthathione-synthase, superoxide-dismutase), but are also responsible for the stimulation of protein mediators of innate pro-survival mechanisms. A further mechanism behind the protective effects of dynamic preservation approaches is the presence of shear stress and as such active perfusion during the preservation phase may induce specific shear stress-sensitive genes some of which include Kruppel-like factor 2 or endothelial nitric oxide synthase. Currently, three multicenter RCTs have completed their patient recruitment and clinical results are expected for the year 2021. The Zurich group initiated a multicentric RCT to assess the impact of HOPE on any DBD liver graft including retransplantations and marginal livers and is powered to assess major complications (Clavien grade ≥III) (NCT01317342). The Groningen team explores the dual HOPE (d-HOPE) technique in DCD grafts (NCT02584283) and our own group initiated a multicentric RCT on HOPE in ECD-DBD liver transplantation in 2017 (NCT03124641).

Viability assessment during MP can guide the clinical decision whether to accept a liver for transplantation and is therefore an important emerging tool in ECD OLT. The possibility of a reliable viability assessment is advocated as a considerable advantage of normothermic perfusion techniques. By sustaining full metabolism, NMP allows to analyse several makers of liver function and injury, including biliary parameters (e.g. bile flow, bile glucose, bicarbonate and pH), perfusate pH and base excess, portal venous- and hepatic artery flow and perfusate hepatocellular enzymes. Despite the reduced metabolic activity during cold storage and hypothermic liver perfusion, there is increasing evidence that a prediction of future graft performance after transplantation may be possible during HOPE, as well. Analysis of the cold perfusate during HOPE provides a unique opportunity to identity potential biomarkers which are associated with various post-OLT outcomes. A recent study involving 31 human ECD-DBD grafts initially rejected for transplantation, found that cold perfusion not only ameliorates reperfusion injury but also allows for graft viability assessment. Thus, the 2-hour perfusate AST and lactate dehydrogenase (LDH) correlated significantly with the peak AST after implantation. In two grafts with a significant postreperfusion transaminase release, a high portal perfusion pressure was noted.

The Zurich group has recently presented a new mitochondrial marker to assess viability of entire liver grafts during HOPE. Real-time fluorometric analysis of mitochondrial flavin mononucleotide (FMN) in the HOPE perfusate predicted human liver function, complications and graft loss prior to transplantation. The use of this surrogate parameter could facilitate proper clinical decision making whether to accept or decline allografts in the HOPE setting. This marker is currently validated in other solid organs and also in the RCT of Guarerras working group. Importantly, the quantification of FMN is possible in real time, requiring only a spectroscope to reliably predict graft survival within the first 30-45 minutes of HOPE. The clinical value and head-to-head comparison of various allograft viability parameters in the HOPE vs. NMP setting has yet to be explored in the setting of a large multicenter RCT. With the advent of clinical MP and the context of a dire donation situation in the western world, it will be of utmost clinical importance to identify the most effective dynamic preservation technique. While past and current clinical trials in DCD and DBD liver transplantation were designed to compare different MP approaches with CCS as the clinical standard, a direct comparison between different end-ischemic MP techniques (HOPE versus NMP) is still lacking.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Patients 18 years or older
* Patients suffering from end stage-liver disease and/or malignant liver tumours
* Listed for OLT
* Receiving ECD-allografts

Exclusion Criteria:

* Recipients of split or living donor liver transplants
* Previous liver transplantation
* Combined transplantations (liver-kidney, liver-lung, etc.)
* Participation in other liver related trials
* The subject received an investigational drug within 30 days prior to inclusion
* The subject is unwilling or unable to follow the procedures outlined in the protocol
* The subject is mentally or legally incapacitated
* Patient is not able to understand the procedures due to language barriers
* Family members of the investigators or employees of the participating departments

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Estimated)
Dates: Start 2021-01-14 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications | After the first 90-days postoperatively
  Comprehensive Complication Index (CCI) (assessed after the first 90-days postoperatively)

SECONDARY OUTCOMES:
Peak alanine aminotransferase (ALT) | During the first week postoperatively
  Peak serum alanine aminotransferase-ALT
Peak aspartate aminotransferase (AST) | During the first week postoperatively
  Peak serum aspartate aminotransferase-AST
Early allograft dysfunction (EAD) | During the first week postoperatively
  Olthoff criteria (bilirubin 10mg/dL on day 7, international normalized ratio 1.6 on day 7, and alanine or aspartate aminotransferases >2000 IU/L)
Primary non-function (PNF) | During the first week postoperatively
  Graft with poor function requiring re-transplantation or leading to death within 7 days after the primary procedure without any identifiable cause of graft failure
Biliary complications | at 6 months postoperatively
  as assessed by MRI / MRCP
Organ utilization rate | During the first week postoperatively
  Rate of donor-allograft offers that result in liver transplantation
Total organ preservation time | Before preservation (HOPE or NPM or CCS), after liver implantation (0-3 hours)
  Organ logistics
Duration and costs of initial intensive care unit (ICU) stay | Subjects will be followed for 6 months postoperatively
  Length of initial Intensive care unit (ICU) stay is determined in days of admission following liver transplantation.
Duration of hospital stay | Subjects will be followed for 6 months postoperatively
  Length of hospital stay is determined in days of hospital admission after discharge and up to six months after liver transplantation
Costs of hospital stay | Subjects will be followed for 6 months postoperatively
  Costs of hospital stay is determined in days of hospital admission after discharge and up to six months after liver transplantation
Postoperative complications | Subjects will be followed for one year postoperatively
  According to the Comprehensive complication index (CCI)
Postoperative major complications | Subjects will be followed for one year postoperatively
  According to the Clavien-Dindo complication score
One-year recipient- and graft survival | Subjects will be followed for one year postoperatively
  One year patient and graft survival

CONTACTS AND LOCATIONS:
Overall Officials: Georg Lurje, M.D., Principal Investigator — Charite University, Berlin, Germany
Locations (4):
- Germany (4):
  - Charité Universitätsmedizin - Berlin, Campus Charité Mitte | Campus Virchow-Klinikum, Berlin
  - University Hospital Bonn, Department of Surgery, Bonn
  - Medizinische Hochschule Hannover (MHH), Department of Surgery and Transplantation, Hanover
  - University Hospital Heidelberg, Department of Surgery and Transplantation, Heidelberg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study webpage — http://www.hopeliver.com